CLINICAL TRIAL: NCT02341144
Title: Percutaneous Rectus Sheath Block Versus Intra-operative Rectus Sheath Block for Pediatric Umbilical Hernia Repair: A Prospective, Randomized Study
Brief Title: Percutaneous Rectus Sheath Block Versus Intra-operative Rectus Sheath Block for Pediatric Umbilical Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00041103
Record Dates: First submitted 2014-12-09; First posted 2015-01-19 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-op percutaneous rectus sheath block (Active Comparator): ultrasound-guided, percutaneous rectus sheath block with ropivacaine by a qualified anesthesiologist
  Interventions: Procedure: Pre-op percutaneous rectus sheath block; Drug: Ropivacaine
- Intra-operative rectus sheath block (Active Comparator): rectus sheath block with ropivacaine under direct visualization by the attending surgeon
  Interventions: Procedure: Intra-operative rectus sheath block; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Pre-op percutaneous rectus sheath block — After induction of anesthesia, the attending anesthesiologist will use a portable ultrasound probe to locate the rectus sheath. A 22 gauge needle will be used to inject a predetermined volume of 0.2% ropivacaine (1cc/kg, max dose 10cc, divided into equal doses bilaterally). The analgesic will be injected percutaneously using ultrasound guidance between the rectus abdominis muscle and the posterior rectus sheath at the lateral border bilaterally.
  Arms: Pre-op percutaneous rectus sheath block
Procedure: Intra-operative rectus sheath block — After the completion of the umbilical hernia repair, after fascial closure, but prior to skin closure, a predetermined volume of 0.2% ropivacaine (1cc/kg, max dose 10c, divided into equal doses bilaterally) will be administered under direct visualization into the rectus sheath bilaterally by the attending surgeon.
  Arms: Intra-operative rectus sheath block
Drug: Ropivacaine
  Other Names: Naropin

SUMMARY:
This is a prospective, double-blinded, randomized controlled study comparing the efficacy of pre-incisional percutaneous rectus sheath block to intra-operative rectus sheath block under direct visualization prior to closure of the incision for providing post-operative analgesia following umbilical hernia repair in children. The current management for reducible umbilical hernias is umbilical hernia repair under general anesthesia as an outpatient procedure.

Patients aged 3-18 years old with a diagnosis of umbilical hernia will be screened for study inclusion. Eligible patients and their parents/guardians will be approached and, if agreeable, consented for the study pre-operatively. Patients will be randomized to receive either pre-incisional percutaneous rectus sheath block by the anesthesiologist or intra-operative rectus sheath block under direct visualization prior to closure of the skin incision by the surgeon. The patient, patient guardians, select research team members, and post-anesthesia care unit (PACU) staff will be blinded to the method of analgesic administration.

DETAILED DESCRIPTION:
Regional anesthesia has been increasingly utilized for providing post-operative analgesia for a number of surgical procedures in children. Rectus sheath block and local anesthetic infiltration of the surgical site are two common modes for providing post-operative analgesia following umbilical hernia repair. Studies comparing the two modes have shown ultrasound-guided rectus sheath block to improve immediate pain scores and reduce use of post-operative analgesia in pediatric patients undergoing umbilical hernia repair. However, these studies have compared pre-incisional ultrasound-guided rectus sheath block to post-operative local anesthetic infiltration as a subcutaneous and/or intradermal injection.

The purpose of the investigators' study is to compare the efficacy of pre-incisional percutaneous rectus sheath block to intra-operative rectus sheath block under direct visualization prior to closure of the skin for providing post-operative analgesia following umbilical hernia repair in children.

The investigators propose a prospective study where pediatric patients who are undergoing elective umbilical hernia repair will be randomized pre-operatively to receive either pre-incisional, ultrasound guided percutaneous rectus sheath block or intra-operative rectus sheath block under direct visualization prior to closure of the skin. The primary outcome is the post-operative pain rating based on the Wong-Baker Faces Pain Rating Scale (WBFPRS) following umbilical hernia repair. Additional outcomes measured will include: operative times, the use of intravenous/oral opioid and/or non-opioid medication in the post-operative period, duration of analgesia following surgery based on time to first rescue analgesic, intra-operative hemodynamic changes, post-operative hemodynamic changes, incidence of side-effects, and complications. Patients/patient guardians will receive a sheet to document post-operative WBFPRS scores, oral opioid and non-opioid medication administration once discharged to home for a total of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3-18 years undergoing elective umbilical hernia repair

Exclusion Criteria:

* Strangulated or incarcerated umbilical hernia (non-elective)
* Allergy to bupivacaine/ropivicaine
* Concurrent surgical procedures
* Developmental delay or neurologic diagnosis that would interfere with post-operative pain score assessment
* Chronic pain medication use
* Chronic pain disorder or complex regional pain syndrome
* Anesthesiologist classification of III or greater.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Chandler, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-op Percutaneous Rectus Sheath Block: ultrasound-guided, percutaneous rectus sheath block by a qualified anesthesiologist
  Pre-op percutaneous rectus sheath block: After induction of anesthesia, the attending anesthesiologist will use a portable ultrasound probe to locate the rectus sheath. A 22 gauge needle will be used to inject a predetermined volume of 0.2% ropivacaine (1cc/kg, max dose 10cc, divided into equal doses bilaterally). The analgesic will be injected percutaneously using ultrasound guidance between the rectus abdominis muscle and the posterior rectus sheath at the lateral border bilaterally.
  Ropivacaine
- Intra-operative Rectus Sheath Block: rectus sheath block under direct visualization by the attending surgeon
  Intra-operative rectus sheath block: After the completion of the umbilical hernia repair, after fascial closure, but prior to skin closure, a predetermined volume of 0.2% ropivacaine (1cc/kg, max dose 10c, divided into equal doses bilaterally) will be administered under direct visualization into the rectus sheath bilaterally by the attending surgeon.
  Ropivacaine
Period: Overall Study
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
Started | 30 | 31
Completed | 28 | 30
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Median (Full Range); unit: years] | 6.2 [3.2 to 15.4] | 6.2 [4.1 to 17.2] | 6.2 [3.2 to 17.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 12 | 13 | 25
Body mass index (BMI) percentile [Median (Full Range); unit: percentile] — body mass index (BMI) percentile: weight (kg) divided by height (m) relative to other children in the US of the same age and sex
  percentile | 57 [3 to 99] | 77 [5 to 98] | 61.2 [3 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain Rating
Description: Using the Wong-Baker FACES Pain Rating Scale (WBFPRS)- pain scores range from zero (no pain) to ten (worst pain) and the average score was reported
Time Frame: from entry in post-anesthesia care unit (PACU) until discharge, estimated 1-2 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
Number analyzed (Participants) | 28 | 30
units on a scale | 2.6 [0 to 6.7] | 3.3 [0 to 8]
Statistical Analysis 1: Comparison: Pre-op Percutaneous Rectus Sheath Block vs Intra-operative Rectus Sheath Block; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to First Narcotic
Description: duration until patient received first dose of narcotic in PACU
Time Frame: from entry in post-anesthesia care unit (PACU) to first narcotic
Measure: Median (Full Range); unit: minutes
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
Number analyzed (Participants) | 28 | 30
minutes | 30 [4 to 54] | 22 [2 to 112]
Statistical Analysis 1: Comparison: Pre-op Percutaneous Rectus Sheath Block vs Intra-operative Rectus Sheath Block; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain Score of Zero
Description: proportion who reported a score of zero throughout their PACU stay using the Wong-Baker (WB) scale with zero being "no pain"
Time Frame: from entry in the post-anesthesia care unit (PACU) until discharge, estimated 1-2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
Number analyzed (Participants) | 28 | 30
Participants | 5 | 3
Statistical Analysis 1: Comparison: Pre-op Percutaneous Rectus Sheath Block vs Intra-operative Rectus Sheath Block; Test type: Superiority; p = 0.39, Chi-squared

4. Secondary Outcome: PACU Morphine Equivalents
Description: morphine equivalents received in PACU
Time Frame: from entry in post-anesthesia care unit (PACU) until discharge, estimated 1-2 hours
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
Number analyzed (Participants) | 28 | 30
mg/kg | 0.04 [0 to 0.24] | 0.09 [0 to 0.2]
Statistical Analysis 1: Comparison: Pre-op Percutaneous Rectus Sheath Block vs Intra-operative Rectus Sheath Block; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: PACU Length of Stay (LOS)
Description: duration of time spent in the post-anesthesia care unit (PACU) from arrival to discharge
Time Frame: from entry in post-anesthesia care unit (PACU) until discharge, estimated 1-2 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
Number analyzed (Participants) | 28 | 30
minutes | 76 [56 to 159] | 80 [49 to 173]
Statistical Analysis 1: Comparison: Pre-op Percutaneous Rectus Sheath Block vs Intra-operative Rectus Sheath Block; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 30 days postoperatively
Arm/Group | Pre-op Percutaneous Rectus Sheath Block | Intra-operative Rectus Sheath Block
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes